CLINICAL TRIAL: NCT02149849
Title: Lateral Surgical Positioning for Thoracic Surgery -Effect on Ipsilateral Shoulder Pain?
Brief Title: Surgical Positioning of the Arm During Thoracic Surgery -Effect on Shoulder Pain After Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Stein Ove Danielsen, RN, MNSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/406
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Ipsilateral shoulder pain; Surgical positioning; Lung cancer; Thoracotomy; Video assisted thoracic surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard lateral positioning (No Intervention)
- Modified lateral positioning (Experimental): Modified lateral positioning. This will ensure less pressure and stretch on shoulder than standard lateral positioning.
  Interventions: Procedure: Modified lateral positioning.

INTERVENTIONS:
Procedure: Modified lateral positioning. — Right before surgery, the patient are posistioned in lateral position with arm elevated (not more than 90 degree from torso). In the intervention, the arm will be lowered and placed in towards the torso for patients enrolled in the experimantal arm.
  Arms: Modified lateral positioning

SUMMARY:
Up to 85% experience shoulder pain after thoracic surgery, especially on the same side as surgery are performed. Referred phrenic nerve pain is probably one cause of ipsilateral shoulder pain (ISP), and positioning of the arm during surgery another. Studies indicates that ISP can be caused by the positioning of the patient during surgery due to muscle -and ligament strain. Can a change in the surgical positioning (less press and stretch) of the ipsilateral arm effect the shoulder pain after thoracic surgery?

ELIGIBILITY:
Inclusion Criteria:

* Men and women;18 years and older
* Thoracotomy for lung cancer
* Video assisted thoracic surgery for lung cancer.

Exclusion Criteria:

* Received treatment for shoulder pain
* Use pain medication on regular basis
* Under 18 year
* Length of stay in ICU more than 24 hours after surgery
* Does not understand the native language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Postoperative shoulder pain after lung surgery. | 3 months
  Using visual analog scale for assesing pain in the shoulder (Scale from 0-10). Mesauring times: VAS pain related to the shoulder before surgery, VAS pain shoulder at day 1 and 3 after surgery. Further will Oslo University Hospital scheme for registration of pain for location and characteristic also be used.

SECONDARY OUTCOMES:
Pain medication | 3 months
  All extra pain medication patient use after surgery until day 4, type and dose, will be mesaured.
White blood cell | 3 months
  Mesaured before surgery, and at day 1 and 3 after surgery.
C reactive protein | 3 months
  Measured before surgery, and at day 1 and 3 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Stein O Danielsen, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway